CLINICAL TRIAL: NCT05243758
Title: The Comparison Of Video Fiberscope And Video Laryngoscope,With Egri Score> 4
Brief Title: Who is Rapid And Success? The Comparison Of Video Fiberscope And Video Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Halil CEBECI, Resident ,Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: B.30.2.ODM.0.20.08/1822
Record Dates: First submitted 2021-12-05; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2018-11

CONDITIONS: Intubation; Difficult or Failed; Airway Responsiveness

STUDY DESIGN:
Intervention Model Description: 60 patients aged between 18-65 years, who were operated in the operating room of our hospital, with an EGRI score of >4 and an ASA (American Society of Anesthesiologists) score of <4 were included.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group video fiberscope of experienced practitioner (Active Comparator): More experienced physician: endotracheal intubation with video fiberscope Assoc. Dr. The group in which Ersin Köksal performed endotracheal intubation using a video fiberscope( Karl Storz GmbH &Co. KG, Tuttlingen, Germany) consisted of 15 patients.Endotracheal intubation was performed by two practitioners using two different devices. Intubation times, number of attempts, failed attempts, postoperative complications and hemodynamic responses were recorded.
  Interventions: Device: Group video fiberscope of experienced practitioner; Device: Group video fiberscope of less experienced practitioner
- Group video laryngoscope of experienced practitioner (Active Comparator): More experienced physician: Endotracheal intubation with DCI video laryngoscopeThe group in which Assoc. Dr. Ersin Köksal performed endotracheal intubation using a DCI video laryngoscope(Storz DCI Video Laryngoscope (Karl Storz GmbH &Co. KG, Tuttlingen, Germany) consisted of 15 patients.Endotracheal intubation was performed by two practitioners using two different devices. Intubation times, number of attempts, failed attempts, postoperative complications and hemodynamic responses were recorded.
  Interventions: Device: Group video laryngoscope of experienced practitioner; Device: Group video laryngoscope of less experienced practitioner
- Group video fiberscope of less experienced practitioner (Active Comparator): Endotracheal intubation with video fiberscope: The group in which DrHalil Cebeci applied endotracheal intubation using a video fiberscope( Karl Storz GmbH &Co. KG, Tuttlingen, Germany) consisted of 15 patients. Endotracheal intubation was performed by two practitioners using two different devices. Intubation times, number of attempts, failed attempts, postoperative complications and hemodynamic responses were recorded.
  Interventions: Device: Group video fiberscope of experienced practitioner; Device: Group video fiberscope of less experienced practitioner
- Group video laryngoscope of less experienced practitioner (Active Comparator): Endotracheal intubation with DCI video laryngoscope:The group in which Dr.Halil Cebeci applied endotracheal intubation using a DCI video laryngoscope(Karl Storz GmbH &Co. KG, Tuttlingen, Germany) consisted of 15 patients.Endotracheal intubation was performed by two practitioners using two different devices. Intubation times, number of attempts, failed attempts, postoperative complications and hemodynamic responses were recorded.
  Interventions: Device: Group video laryngoscope of experienced practitioner; Device: Group video laryngoscope of less experienced practitioner

INTERVENTIONS:
Device: Group video fiberscope of experienced practitioner — One of the classical alternatives to laryngoscopy in difficult endotracheal intubation is video laryngoscopyvideo fiberscope( Karl Storz GmbH &Co. KG, Tuttlingen, Germany). Reaching the image from the patient with pre- and from the cervical point of view, or from the cervical point of view, to be completed with a good view from a large screen to be completed with an image before and within intubation. It also facilitates learning in education.
  Arms: Group video fiberscope of experienced practitioner; Group video fiberscope of less experienced practitioner
Device: Group video laryngoscope of experienced practitioner — Intubation Pending Difficult as well as challenging . Fiberoptic (fiberscope) intubation is the gold standard in difficult airway. Lacking this supplement, it will be widely used for practice, as it is suitable for video laryngeal.
  Arms: Group video laryngoscope of experienced practitioner; Group video laryngoscope of less experienced practitioner
Device: Group video fiberscope of less experienced practitioner — One of the classical alternatives to laryngoscopy in difficult endotracheal intubation is video laryngoscopy video fiberscope( Karl Storz GmbH &Co. KG, Tuttlingen, Germany). Reaching the image from the patient with pre- and from the cervical point of view, or from the cervical point of view, to be completed with a good view from a large screen to be completed with an image before and within intubation. It also facilitates learning in education.
  Arms: Group video fiberscope of experienced practitioner; Group video fiberscope of less experienced practitioner
Device: Group video laryngoscope of less experienced practitioner — Entubation pending difficult as well as challenging . Fiberoptic (fiberscope) intubation is the gold standard in difficult airway. Lacking this supplement, it will be widely used for practice, as it is suitable for video laryngeal.Storz DCI Video Laryngoscope (Karl Storz GmbH &Co. KG, Tuttlingen, Germany)
  Arms: Group video laryngoscope of experienced practitioner; Group video laryngoscope of less experienced practitioner

SUMMARY:
Endotracheal intubation plays an important role in general anesthesia. Complications can be prevented by using alternative airway devices in predetermined difficult intubation cases. In this study, the investigators aimed to compare the results of endotracheal intubation with video fiberscope and DCI video laryngoscope devices of two different experienced physicians (E and H).

DETAILED DESCRIPTION:
In this randomized and prospective study, 60 patients with EGRI score> 4 and ASA score <4, operated between 1 October 2018 and 1 March 2019 in Ondokuz Mayıs University Medical Faculty Hospital were included. Endotracheal intubation was performed by two practitioners using two different devices. Intubation times, number of attempts, failed attempts, postoperative complications and hemodynamic responses were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Operated in the operating room of our hospital,
* Aged 18-65,
* EGRI score>4,
* ASA (American Society of Anesthesiologists) score<4

Exclusion Criteria:

* Cerebrovascular disease (cerebral ischemia, hemorrhage or stroke), presence of carotid stenosis or history of coronary artery disease,

  * Neurological disorders (history of chronic headache, epilepsy or head trauma), alcohol or psychoactive drug addiction,
  * Serious heart and/or lung diseases, liver and/or kidney failure,
  * Uncontrolled diabetes and/or hypertension,
  * Dental abscess,
  * Mouth opening <1.5 cm,
  * Known bleeding disorder,
  * Pregnancy,
  * Mental retardation,
  * Contraindications to drugs, allergy to drugs used,
  * Patient rejection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Intubation times, | during intubation
  The moment when the endotracheal intubation tube was passed between the vocal cords following the vocal cord image obtained with the device was recorded in seconds. In endotracheal intubation performed with a video fiberscope, the end of the fiberscope with a camera passing through the vocal cords, and in endotracheal intubation performed with a DCI video laryngoscope, the intubation tube passing between the vocal cords was counted as successful intubation time.
Number of attempts | during intubation for patients,
  The procedure will be considered unsuccessful if intubation is unsuccessful in three attempts, if the intubation process exceeds three minutes, or if the peripheral oxygen saturation (SpO2) is <90% during this period. If this situation was encountered, it was planned to ventilate the patient with an anesthesia mask until the oxygen saturation approached 100% and to use alternative airway devices.
Time to find the glottis: | during intubation for patients
  The time from the moment the device entered between the patient's anterior incisors until the vocal cords were seen was recorded in seconds.
Blood pressure | During intubation, at 1st, 2nd and 5th minutes after intubation
  Hemodynamic parameters; heart rate (/min), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), mean arterial pressure (mmHg), and SpO2 were recorded before induction (baseline), during intubation, at 1st, 2nd and 5th minutes after intubation
Pulse oximeter | Before induction (baseline), during intubation, at 1st, 2nd and 5th minutes after intubation
  Oximetry is a convenient and painless alternative to needlesticks, is simple to use, and provides immediate data. These advantages make oximetry an invaluable tool for determination the client's need for oxygen therapy and assessing effectiveness of therapy. The oximeter registers arterial oxygen saturation (SaO2). An SaO2 greater than 95% is considered normal, whereas values lower than 93% usually indicate the need for oxygen therapy and further assessment.

CONTACTS AND LOCATIONS:
Overall Officials: ERSIN KOKSAL, PROFFOSOR, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University Faculty of Medicine, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No